CLINICAL TRIAL: NCT00398489
Title: Evaluation of Response Rate to Pre-Operative Docetaxel + Herceptin Study Part A and Docetaxel Study Part B in Locally Advanced Breast Cancer Patients, Stratified by HER2-Status Trial - PHASE II [(Herceptin Docetaxel Neoadjuvant) HEDON]
Brief Title: Docetaxel, Epirubicin, and Cyclophosphamide With or Without Trastuzumab in Treating Women With Locally Advanced Breast Cancer That Can Be Removed By Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000516034; KRDI-TUM-HED-324-PAE-0090-I; EU-20634; EUDRACT-2005-000967-24
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage II breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab; Anastrozole; Cyclophosphamide; Docetaxel; Epirubicin; Goserelin; Tamoxifen; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Biological: trastuzumab
Drug: anastrozole
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: goserelin acetate
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, epirubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy with or without monoclonal antibody therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving docetaxel, epirubicin, and cyclophosphamide with or without trastuzumab works in treating women with locally advanced breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of neoadjuvant therapy comprising docetaxel and trastuzumab (Herceptin®) and adjuvant therapy comprising epirubicin hydrochloride, cyclophosphamide, and trastuzumab (Herceptin®) followed by radiotherapy in women with locally advanced, HER2-positive, operable breast cancer.
* Determine the efficacy of neoadjuvant therapy with docetaxel and adjuvant therapy comprising epirubicin hydrochloride and cyclophosphamide followed by radiotherapy in women with locally advanced, HER2-negative, operable breast cancer.

OUTLINE: This is an open-label, prospective, multicenter study. Patients are stratified according to HER2 status (positive vs negative).

* Neoadjuvant therapy:

  * Stratum 1 (HER2-positive disease): Patients receive trastuzumab IV over 30-90 minutes on days 1, 8, and 15 and docetaxel IV over 60 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity
  * Stratum 2 (HER2-negative disease): Patients receive docetaxel IV alone as in stratum 1.
* Surgery: All patients undergo surgery in week 19.
* Adjuvant therapy: Beginning within 2 weeks after surgery, patients receive adjuvant therapy.

  * Stratum 1 (HER2-positive disease): Patients receive trastuzumab IV over 30-90 minutes on days 1, 8, and 15, epirubicin hydrochloride IV over 30 minutes on day 2, and cyclophosphamide IV over 30 minutes on day 2. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV alone every 3 weeks until week 52.
  * Stratum 2 (HER2-negative disease): Patients receive epirubicin hydrochloride and cyclophosphamide as in stratum 1.
* Radiotherapy: Patients who undergo breast conserving surgery or patients who undergo mastectomy with ypN positive lymph nodes (i.e., > 4 positive lymph nodes) or ypT3 tumor (i.e., tumor size > 4 cm) undergo radiotherapy, beginning in approximately week 31 and continuing until up to week 38.
* Adjuvant endocrine therapy: Patients with estrogen receptor- or progesterone receptor-positive disease receive adjuvant endocrine therapy beginning in approximately week 31. Premenopausal patients ≤ 40 years of age receive goserelin for 2-3 years and tamoxifen citrate for 5 years.Premenopausal patients > 40 years of age receive tamoxifen citrate for 5 years. Postmenopausal patients receive anastrozole for 5 years years.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 94 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary carcinoma of the breast by core biopsy
* Solitaire or multifocal disease, defined as tumor manifestations within a quadrant or distance between tumor manifestations measured bilaterally < 4 cm, respectively

  * No multifocal primary tumor, defined as tumor manifestations in different quadrants or distance between tumor manifestations ≥ 4 cm
* Locally advanced, operable disease

  * Primary tumor ≥ 2 cm by clinical examination or imaging (i.e., mammogram, MRI, or ultrasound)

    * Inflammatory breast cancer with bidimensionally measurable lesion, independent of nodal status, allowed
* HER2 status meeting 1 of the following criteria:

  * HER2-positive disease

    * 3+ by immunohistochemistry (IHC) and/or positive by fluorescence in situ hybridization (FISH)
  * HER-2 negative disease

    * 0 or 1+ by IHC OR 2+ by IHC and negative by FISH
* No distant metastases by clinical or imaging diagnosis
* No prior breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Pre- or post-menopausal
* ECOG performance status 0-2
* Platelet count ≥ 100,000/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 10 g/dL
* ALT and AST ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Bilirubin normal (unless due to clearly documented Gilbert's syndrome)
* Not pregnant or nursing
* Negative pregnancy test (for premenopausal women or women with a postmenopausal status for < 1 year)
* Fertile patients must use effective contraception
* Adequate organ function for cytotoxic chemotherapy
* No known hypersensitivity reaction to the study agents or incorporated substances
* No known allergy or severe reactions to trastuzumab or its constituents (for patients with HER2-positive disease)
* No preexisting motor or sensory neuropathy ≥ grade 2
* No other invasive malignancy within the past 5 years that would preclude study compliance or affect the interpretation of study results
* LVEF ≥ 55% by MUGA or echocardiography
* No other serious illness or medical condition, including any of the following:

  * New York Heart Association class II-IV congestive heart failure
  * History of documented congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction within the past 12 months
  * Uncontrolled hypertension (i.e., systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg)
  * Clinically significant valvular heart disease
  * High-risk, uncontrolled arrhythmias
  * Dyspnea at rest due to malignant or other disease
  * Condition that requires supportive oxygen therapy
  * Active serious uncontrolled infections
  * Uncontrolled diabetes

PRIOR CONCURRENT THERAPY:

* No prior systemic therapy for cancer
* No prior trastuzumab (Herceptin^®) (for HER2-positive patients)
* No other concurrent anticancer therapy
* No other concurrent investigational drugs
* No concurrent immunosuppressive therapy
* No concurrent sex hormones
* No concurrent corticosteroids unless for premedication
* No concurrent bisphosphonates during active treatment with chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Rate of pathologic complete remission (pCR) after neoadjuvant therapy comprising docetaxel and trastuzumab (Herceptin®) in women with locally advanced, HER2-positive, operable breast cancer
Rate of pCR after neoadjuvant docetaxel in women with locally advanced, HER2-negative, operable breast cancer
Tolerability of treatment as measured by the nature and frequency of adverse events in women with HER2-positive or HER2-negative disease
Identification of predictive markers

SECONDARY OUTCOMES:
Rate of breast conserving therapy versus mastectomy in comparison to preoperative evaluation
Correlation of clinical/sonographical response with pathological response, including lymph node status
Rate of clinical complete remission (cCR) after neoadjuvant therapy comprising docetaxel and trastuzumab in women with locally advanced, HER2-positive, operable breast cancer
Rate of cCR after neoadjuvant docetaxel in women with locally advanced, HER2-negative, operable breast cancer
Disease-free survival after 2.5 and 5 years
Overall-survival after 2.5 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Paepke, MD, Study Chair — Technical University of Munich
Locations (5):
- Germany (5):
  - Klinikum Bayreuth, Bayreuth
  - Universitaetsfrauenklinik - Koeln, Cologne
  - Klinikum Deggendorf, Deggendorf
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich